CLINICAL TRIAL: NCT03607383
Title: Red Rice Yeast in Low-density Lipoprotein (LDL) Lowering: an Efficacy Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRY2018
Record Dates: First submitted 2018-06-26; First posted 2018-07-31 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Dyslipidemias; LDL Hyperlipoproteinemia
Keywords: statins; red rice yeast; adverse effects; cholesterol, LDL; treatment outcome; tolerability
MeSH Terms: conditions — Dyslipidemias | interventions — red yeast rice; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Red rice yeast group (Experimental): Red rice yeast based product will be provided under the brand name Molval Fort, one pill a day, for 8 weeks, for a moderate intensity treatment equivalent according the American College of Cardiology/American Heart Association (ACC/AHA) guidelines definitions
  Interventions: Drug: Red Rice Yeast Extract
- Statin group (Active Comparator): Statin choice is done at the discretion of the treating physician for a moderate intensity treatment equivalent according the American College of Cardiology/American Heart Association (ACC/AHA) guidelines definitions, for 8 weeks
  Interventions: Drug: Statin

INTERVENTIONS:
Drug: Red Rice Yeast Extract — adults requiring moderate intensity treatment will be provided red rice yeast extracts or statins, depending on the randomization; followed for compliance and adverse effects check, and reevaluated in a final visit with blood test after 8 weeks
  Arms: Red rice yeast group
Drug: Statin — Statin choice is done at the discretion of the treating physician for a moderate intensity treatment equivalent according the American College of Cardiology/American Heart Association (ACC/AHA) guidelines definitions, for 8 weeks
  Arms: Statin group

SUMMARY:
Red yeast rice is a source of active compounds in reducing LDL levels with practically no side effects. Molval Fort is a natural product available in the Lebanese market with a combination of red yeast rice extracts, EPA/DHA and coenzyme Q10.

The investigators are conducting this study to explore the effect of red yest rice extracts based product on LDL and its side effects in a sample of primary care Lebanese patients.

DETAILED DESCRIPTION:
Red yeast rice is a source of active compounds in reducing LDL levels with practically no side effects. Studies performed on American and Chinese populations have shown positive results. These studies need confirmation in different populations. Molval Fort is a natural product available in the Lebanese market with a combination of red yeast rice extracts, EPA/DHA and coenzyme Q10. The investigators are conducting this study to explore the effect of red yest rice extracts based product on LDL and its side effects in a sample of primary care Lebanese patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>18 years)
* Indication to mild or moderate statin based on AHA 2013 guidelines
* Treatment naïve

Exclusion Criteria:

* Allergy to rice
* Renal or hepatic terminal disease
* Any contra indication to statin treatment
* Pregnancy wish during study period
* Familial hypercholesterolemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-02-07 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
LDL reduction | eight weeks
  after an eight week treatment, cholesterol LDL levels' reduction is compared in the two groups

SECONDARY OUTCOMES:
incidence of side effects | eight weeks
  after eight weeks of treatment, the incidence of side effects is studied among the red rice yeast group

OTHER OUTCOMES:
physician and patient satisfaction | eight weeks
  physician and patient satisfaction will be evaluated by a single question questionnaire: Were you satisfied by the treatment?

CONTACTS AND LOCATIONS:
Overall Officials: Marouan Zoghbi, Principal Investigator — Hôtel Dieu de France Hospital
Locations (1):
- Saint Anthony Primary Care Center, Jdeïdé, Lebanon

IPD SHARING:
Plan to Share IPD: No